CLINICAL TRIAL: NCT06253624
Title: Gait Pattern Analysis After All Arthroscopic ATFL Repair Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, İnci Hazal Ayas, Research asistant, Gazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Iayas6
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Ankle Lateral Ligament; Gait Analysis
Keywords: ATFL repair; Arthroscopy; Pedobarography; Plantar pressure distribution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATFL surgery (Other): All participants will undergo all arthroscopic ATFL repair surgery.
  Interventions: Procedure: All Arthroscopic ATFL Repair Surgery

INTERVENTIONS:
Procedure: All Arthroscopic ATFL Repair Surgery — The patients undergo surgery with spinal block, general anesthesia, or a combination of both. During the diagnostic arthroscopy, the anterior compartment is examined with a 4 mm 30-degree camera, and lateral ankle instability is diagnosed arthroscopically

SUMMARY:
The study will investigate alterations in post-surgical gait patterns among patients who have undergone all arthroscopic repair surgery for the anterior talofibular ligament (ATFL) due to ankle instability. The gait biomechanics of patients scheduled for surgery will be assessed preoperatively using pedobarographic analysis. Subsequent changes in walking biomechanics will be evaluated and interpreted at the 3rd and 6th postoperative months. Consequently, the impact of the all arthroscopic anatomical ATFL repair method on walking will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Presence of unilateral ankle instability.
* Planning for all arthroscopic anterior talofibular ligament (ATFL) repair surgery.

Exclusion Criteria:

* Presence of foot and ankle deformities.
* Presence of orthopedic or neurological pathologies that may affect walking biomechanics.
* History of prior foot and ankle surgery.
* Assessment of surgical stability deemed unsuccessful at the 3rd or 6th month postoperative control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Pedobarography | one day before surgery
  Pedobarographic analysis involves the completion of the platform, pressure sensors, software, and computer installation for gait analysis.
  In dynamic analysis, the patient takes a step on the platform at a regular walking speed, with arms relaxed at the sides of the body, following a natural gait. In static analysis, measurements are taken while the patient remains stationary on the platform with arms in a free position next to the body. Five measurements are separately recorded for both feet during the step, heel strike, and toe lift phases. These measurements capture the highest pressures on the back of the foot, the middle part of the foot, the inner, middle, lateral side of the front of the foot, and the toes.
  The plantar pressure distribution obtained from the measurement is divided into desired areas (masks). The pressure, force, and pressure-time integral corresponding to each area are then used to determine how and for how long these areas are exposed to pressure.
Pedobarography | 3 months after the surgery
  Pedobarographic analysis involves the completion of the platform, pressure sensors, software, and computer installation for gait analysis.
  In dynamic analysis, the patient takes a step on the platform at a regular walking speed, with arms relaxed at the sides of the body, following a natural gait. In static analysis, measurements are taken while the patient remains stationary on the platform with arms in a free position next to the body. Five measurements are separately recorded for both feet during the step, heel strike, and toe lift phases. These measurements capture the highest pressures on the back of the foot, the middle part of the foot, the inner, middle, lateral side of the front of the foot, and the toes.
  The plantar pressure distribution obtained from the measurement is divided into desired areas (masks). The pressure, force, and pressure-time integral corresponding to each area are then used to determine how and for how long these areas are exposed to pressure.
Pedobarography | 6 months after the surgery
  Pedobarographic analysis involves the completion of the platform, pressure sensors, software, and computer installation for gait analysis.
  In dynamic analysis, the patient takes a step on the platform at a regular walking speed, with arms relaxed at the sides of the body, following a natural gait. In static analysis, measurements are taken while the patient remains stationary on the platform with arms in a free position next to the body. Five measurements are separately recorded for both feet during the step, heel strike, and toe lift phases. These measurements capture the highest pressures on the back of the foot, the middle part of the foot, the inner, middle, lateral side of the front of the foot, and the toes.
  The plantar pressure distribution obtained from the measurement is divided into desired areas (masks). The pressure, force, and pressure-time integral corresponding to each area are then used to determine how and for how long these areas are exposed to pressure.

SECONDARY OUTCOMES:
American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS) | one day before surgery
  The hindfoot score comprises nine questions that assess pain, function, and alignment. Within the survey, one question pertains to pain, seven questions address function, and one question relates to alignment. The pain section is appraised on a scale of 40 points, the function section on 50 points, and the alignment section on 10 points, summing up to a total of 100 points. A higher score indicates better functionality.
American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS) | 3 months after the surgery
  The hindfoot score comprises nine questions that assess pain, function, and alignment. Within the survey, one question pertains to pain, seven questions address function, and one question relates to alignment. The pain section is appraised on a scale of 40 points, the function section on 50 points, and the alignment section on 10 points, summing up to a total of 100 points. A higher score indicates better functionality.
American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS) | 6 months after the surgery
  The hindfoot score comprises nine questions that assess pain, function, and alignment. Within the survey, one question pertains to pain, seven questions address function, and one question relates to alignment. The pain section is appraised on a scale of 40 points, the function section on 50 points, and the alignment section on 10 points, summing up to a total of 100 points. A higher score indicates better functionality.

CONTACTS AND LOCATIONS:
Overall Officials: Ulunay Kanatlı, Study Chair — Gazi University; Mehmet A Tokgöz, Study Director — Gazi University; Zeynep Hazar, Study Director — Gazi University
Locations (1):
- Gazi University Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No